CLINICAL TRIAL: NCT03542903
Title: Clinical Trial Comparing Two Electroconvulsive Therapy (ECT) Application Schemas in Ultra-resistant Schizophrenia
Brief Title: ECT in Ultra-resistant Schizophrenia
Acronym: SURECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier du Rouvray (Other Government)
Collaborators: University Hospital, Rouen (Other); University Hospital, Bordeaux (Other); Nantes University Hospital (Other); University Hospital, Toulouse (Other); University Hospital, Caen (Other); Centre Hospitalier Henri Laborit (Other); Centre Hospitalier St Anne (Other); Centre Hospitalier de Cadillac (Other); Hôpital Louis Mourier (Other); University Hospital, Montpellier (Other); University Hospital, Clermont-Ferrand (Other); Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-A02657-46
Record Dates: First submitted 2018-04-11; First posted 2018-05-31 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia; Electroconvulsive Therapy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: A multicentric, prospective, random-assignment study incorporating both non-blinded treatment and blinded assessment
Who Masked: Outcomes Assessor
Masking Description: non-blinded treatment and blinded assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short ECT arm (Active Comparator): In the short arm, bitemporal ECT is administered twice a week during the first 6 weeks. Afterwards, it is administered once a week during 4 weeks. After that, the patients will have one ECT every 3 weeks during 6 weeks. Lastly, patients will receive one ECT each month during 2 months.
  Interventions: Device: Electroconvulsive therapy
- Long ECT arm (Active Comparator): In the long arm, bitemporal ECT is administered twice a week during the first 12 weeks. Afterwards, it is administered once a week during 8 weeks. After that, the patients will have one ECT every 3 weeks during 12 weeks. Lastly, patients will receive one ECT each month during 4 months.
  Interventions: Device: Electroconvulsive therapy

INTERVENTIONS:
Device: Electroconvulsive therapy — Electroconvulsive therapy is administered through electrodes positioned bilaterally (for quicker efficacy) on the frontotemporal region.
  The stimulation dose is determined by titration method, during the first ECT session.
  The dose for therapeutic stimulation will be twice the seizure threshold. This dose may be increased as the crisis does not meet the effectiveness criteria, as is recommended.
  For patients undergoing ECT, an intravenous injection of etomidate (between 0.1 and 0.7 mg/kg) and suxamethonium chloride (0.8 and 1.2 mg/kg) is performed. The required doses are adapted according to each patient by the anaesthetist and they are documented in the patients' files. A mixture of etomidate and propofol can be used in second-line or just propofol in third-line (no more than 2mg/kg).

SUMMARY:
The effects of the ECT in schizophrenia ultra-resistant were studied in short times (4-6 months in most studies with follow-up). The literature identified a high relapse rate of 32% in the weeks to months after ECT discontinuation. The use of the ECT in the prevention of the relapse is partially known. In an empirical way, experts recommend protocols of prevention of the relapse going from 6 to 12 months. Nevertheless, the profit of a long cure (12 months) compared with a short cure (6 months) was never determined. Therefore, the investigators decided to lead a prospective randomized controlled study in order to compare the response rates between the two strategies of clozapine and ECT combinations applied to URS patients. The treatment consisted either in a short therapy of six months or a longer course of therapy of twelve months. To the investigators' knowledge, it is the first study which compares two ECT strategies (both the short duration and the longer one) for the treatment of URS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with URS: patients who continue to experience persistent positive psychotic symptoms: item score of 4 (moderate) on at least two of four positive symptoms on the BPRS (grandiosity, suspiciousness, hallucinations and unusual thoughts), current presence of at least moderately severe illness on the total BPRS-18 (45) and a score of 4 (moderate) on the CGI-S, despite a period of clozapine therapy of at least 6 weeks with a plasma concentration of 350 ng/ml and at least two unsuccessful previous treatment trials with conventional or atypical antipsychotic drugs from two distinct families at a dose 600 mg of chlorpromazine equivalents.
* Age: from 18 to 55
* Patients with stable treatments for at least 8 weeks (antipsychotics, mood stabilizers and antidepressants).
* Participants who gave their informed, written consents and agreement of their guardian for the patients under guardianship
* Patients deprived of liberty if they gave their informed, written consents

Exclusion Criteria:

* Current affective episode according to DSM-5 criteria;
* ECT within (the last) 6 months;
* Unstable epilepsy ; severe neurological or systemic disorder that could significantly affect cognition, behavior, or mental status (other than late dyskinesia or neuroleptic-induced parkinsonism);
* Severe substance use disorders (other than nicotine or caffeine) according to DSM-5 criteria.
* Concomitant use of antiepileptics and benzodiazepines apart from lamotrigine
* Women of childbearing age with no adequate contraception, pregnant or lactating women;
* Patients having contraindications to etomidate or any of its excipients;
* Patients having contraindications to neuromuscular blocking agents;
* Patients participating or having participated in an interventional clinical trial within 30 days prior to the inclusion visit;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2023-10-04 (Estimated); Study Completion 2023-10-04 (Estimated)

PRIMARY OUTCOMES:
The response rate (a 30% decrease in the Positive and Negative Syndrome Scale (PANSS)) at 15th month | three months after the end of the treatment (i.e. 9 and 15 months)
  The response rate (a 30% decrease in the PANSS, ranging from 30, the minimum, to 210, the most severe score) at 15th month

SECONDARY OUTCOMES:
The response rate (a 30% decrease in the Brief Psychiatric Rating Scale (BPRS)) | three months after the end of the treatment (i.e. 9 and 15 months)
  The response rate (a 30% decrease in the BPRS, ranging from 18, the minimum, to 126, the most severe score) at 15th month.
The response rate (a 30% decrease in the BPRS) at different times of the study | 2, 4, 6 and 12 months
  The response rate (a 30 % decrease in the BPRS) at 2, 4, 6 and 12 months.
Response rate (a 30% decrease in the PANSS) at different times of the study | 2, 4, 6 and 12 months
  The response rate (a 30 % decrease in the PANSS) at 2, 4, 6 and 12 months.
Neuropsychological assessment- MMSE | -1, 6 and 15 months
  The scores and variations of the Mini Mental Status Examination (MMSE) at -1, 6 and 15 months.
Neuropsychological assessment- SSTICS | -1, 6 and 15 months
  The scores and variations of the Subjective Scale To Investigate Cognition In Schizophrenia (SSTICS, scores ranging from 0 to 84, the most severe score) at -1, 6 and 15 months.
Neuropsychological assessment- Grober and Buschke test | -1, 6 and 15 months
  The scores and variations of the test of Grober and Buschke at -1, 6 and 15 months.
Neuropsychological assessment- test of doors | -1, 6 and 15 months
  The scores and variations of the test of doors at -1, 6 and 15 months.
Neuropsychological assessment- test of d2 | -1, 6 and 15 months
  The scores and variations of the test of d2 at -1, 6 and 15 months.
Neuropsychological assessment - "figure de Rey" test | -1, 6 and 15 months
  the scores ans variations of the test of " figure de Rey" at -1, 6 and 15 months.
Other clinical assessment- HAMD-21 | day 1 and 2, 4, 6, 9, 12 and 15 months
  The scores and variations of the Hamilton Rating Scale-21 items (HAMD-21, scores ranging from 0 to 64, the most severe score) at day 1 and 2, 4, 6, 9, 12 and 15 months.
Other clinical assessment-YMRS | day 1 and 2, 4, 6, 9, 12 and 15 months
  The scores and variations of the Young Mania Rating Scale (YMRS, scores ranging from 0 to 60, the most severe score) at day 1 and 2, 4, 6, 9, 12 and 15 months.
Other clinical assessment-GAF | day 1 and 2, 4, 6, 9, 12 and 15 months
  The scores and variations of the Global Assessment Functioning (GAF, scores ranging from 0 to 100, the best score) at day 1 and 2, 4, 6, 9, 12 and 15 months.
Other clinical assessment-MOAS | day 1 and 2, 4, 6, 9, 12 and 15 months
  The scores and variations of the Modified Overt Aggression Scale (MOAS, scores ranging from 0 to 100, the most severe score) at day 1 and 2, 4, 6, 9, 12 and 15 months.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Centre Hospitalier Charles Perrens, Bordeaux
  - Centre Hospitalier de Cadillac, Cadillac
  - CHU de Caen, Caen
  - Clermont-Ferrand Hospital, Clermont-Ferrand
  - Montpellier University Hospital, Montpellier
  - CHU de Nantes, Nantes
  - EPS Ville Evrard, Neuilly-sur-Marne
  - Centre Hospitalier Saint Anne, Paris
  - Centre Hospitalier Henri Laborit, Poitiers
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moulier V, Krir MW, Dalmont M; SURECT Group; Guillin O, Rotharmel M. A prospective multicenter assessor-blinded randomized controlled study to compare the efficacy of short versus long protocols of electroconvulsive therapy as an augmentation strategy to clozapine in patients with ultra-resistant schizophrenia (SURECT study). Trials. 2021 Apr 15;22(1):284. doi: 10.1186/s13063-021-05227-3. PMID 33858488